CLINICAL TRIAL: NCT02996370
Title: Effect of I-Shape Incısıon Technique on Inter-Implant Papilla: A Prospective Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Özge PEHLİVANOĞLU, Özge PEHLİVANOĞLU, PhD,DDS Ege University, School of Dentistry, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EGE-OP 2013
Record Dates: First submitted 2016-12-08; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Tooth Loss; Bone Loss
Keywords: esthetic; inter-implant papilla; soft tissue tickness; crestal bone loss; second stage surgery
MeSH Terms: conditions — Tooth Loss; Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group- ı shape incision (Active Comparator): Second stage surgery was made I shape incision technique .
  Interventions: Other: papilla fill index; Other: crestal bone loss; Other: probing depth; Other: Modified sulcus bleeding index; Other: Modified plaque index
- Control group- midcrestal incision (Active Comparator): In the control group second stage surgery was made using the conventional method, midcrestal technique.
  Interventions: Other: papilla fill index; Other: crestal bone loss; Other: probing depth; Other: Modified sulcus bleeding index; Other: Modified plaque index

INTERVENTIONS:
Other: papilla fill index — The clinical photographs were taken baseline, 3 and 6 month. Two T shaped full-round hexagonal straight filaments, each 5 mm, were used in the taking of standardized images.
Other: crestal bone loss — Crestal bone loss was measured on digital radiographs at baseline, 3 and 6 month with a Java program me (Image-J 3.0 NIH, Bethesda, USA)
Other: probing depth — The change of probing depth between baseline, 3 and 6month. Probing depth was measured with a plastic periodontal probe (mm)
Other: Modified sulcus bleeding index — Modified bleeding index was measured baseline, 3 and 6 month. Presence of bleeding on probing were performed at four sites of implants.
Other: Modified plaque index — Modified plaque index was measured baseline, 3 and 6 month. Presence of plaque index was performed at four sites of implants.

SUMMARY:
Regenerating a predictable inter-implant papilla is the most complex and challenging aspect of implant dentistry. The aim of the study was to compare the efficacy of I shaped incision technique and conventional midcrestal incision technique for interimplant papilla reconstruction in a 6 month clinical trial.

DETAILED DESCRIPTION:
A total of 40 implants were placed in 12 patients. Groups were determined at second stage surgery, I shape technique used in test group and mid-crestal technique used in control group. The clinical parameters, including modified plaque index, modified sulcus bleeding index, probing depth, keratinized tissue level were recorded baseline, 3 and 6 month. The vertical distance between the crests top-contact point was evaluated with digital periapical radiographs at baseline 3 and 6 month. Also the clinical photographs were taken baseline, 3 and 6 month. Two T shaped full-round hexagonal straight filaments, each 5 mm, were used in the taking of standardized images. With these images the ratio of the papilla area in proportion to the embrasure area and the papilla classification was measured. Non-parametric test were used for statistically analysis.

ELIGIBILITY:
Inclusion Criteria:

* No sistemic condition, and age > 18 years,
* healthy soft tissue (bleeding on probing (BOP) ≤ 20%, Plaque Index ≤ 15%,
* in a need of at least two collateral implants in the maxilla from second premolar to second premolar
* sufficient keratinized tissue
* no bone augmentation procedures before implant placement
* use of tobacco 10N ≥ cigarettes daily
* sufficient distance between opposite occluding dentition at the proposed implant sites

Exclusion Criteria:

* history of aggressive periodontitis,
* systemic diseases such as diabetes
* pregnant or lactating women
* radiation therapy in the head and neck area wihtin the previous 12 months,
* heavy smokers
* bruxism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
papilla fill index | baseline
  Baseline will be 1 week after cementation of the crowns.
papilla fill index | 3 month
  Papilla fill index will be recorded 3rd month after baseline
papilla fill index | 6 month
  Papilla fill index will be recorded 6th month after baseline
crestal bone loss | Change from baseline crestal bone level up to 3 months
  Crestal bone loss was measured on radiographs between baseline-3rd month.
crestal bone loss | Change from baseline crestal bone level up to 6 months
  Crestal bone loss was measured on radiographs between baseline-6th month.
vertical distance | baseline, 3 and 6 month
  Inter-implant vertical distance between the crests top-contact point was also evaluated with digital periapical radiographs.

SECONDARY OUTCOMES:
Probing depth | baseline
  The level of probing depth at baseline. Probing depth was measured with a plastic periodontal probe.
Probing depth | 3 month
  The level of probing depth at 3 month. Probing depth was measured with a plastic periodontal probe.
Probing depth | 6 month
  The level of probing depth at 6 month. Probing depth was measured with a plastic periodontal probe.
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at baseline
  Modified sulcus bleeding index was recorded at four sites of implants after 10 sec. of probing.
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at 3 month
  Modified sulcus bleeding index was recorded at four sites of implants after 10 sec. of probing.
Modified sulcus bleeding index | Modified sulcus bleeding index was recorded at 6 month
  Modified sulcus bleeding index was recorded at four sites of implants after 10 sec. of probing.
Modified plaque index | Modified plaque index was recorded at baseline
  The dichotomous presence of supra gingival plaque was recorded at four sites of implants
Modified plaque index | Modified plaque index was recorded at 3 month
  The dichotomous presence of supra gingival plaque was recorded at four sites of implants
Modified plaque index | Modified plaque index was recorded at 6 month
  The dichotomous presence of supra gingival plaque was recorded at four sites of implants
Keratinized tissue level | Keratinized tissue level was recorded at baseline
  Keratinized tissue level measured with a plastic periodontal probe
Keratinized tissue level | Keratinized tissue level was recorded at 3 month
  Keratinized tissue level measured with a plastic periodontal probe
Keratinized tissue level | Keratinized tissue level was recorded at 6 month
  Keratinized tissue level measured with a plastic periodontal probe

IPD SHARING:
Plan to Share IPD: Undecided